CLINICAL TRIAL: NCT05756673
Title: Six Month Clinical Efficacy of Virtually Supervised Mouthwash and Interdental Brushes: Effect on Plaque, Gingivitis and Oral Microbiome
Brief Title: A Study of Virtually Supervised Mouthwash and Interdental Brushes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CCSORC004843; CCSORC004843 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2023-02-07; First posted 2023-03-06 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Brush Only (Other): Participants will brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protections Toothpaste for 2 timed minutes under virtual supervision in the morning. At home, participants will brush a second time unsupervised daily in the evening and twice daily over weekends and holidays for the first 3 months of the study (up to visit 3). After visit 3, for the next three months until the end of the study, weekday virtual visits will drop to three times a week. First product use will occur at the site under supervision. Participants will be required to record their daily product use times on a participant diary.
  Interventions: Drug: Colgate Cavity Protection Toothpaste
- Brush/Rinse (LISTERINE ZERO Alcohol Mouthwash COOL MINT) (Experimental): Participants will brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protections Toothpaste for 2 timed minutes and then rinse for 30 seconds with LISTERINE ZERO Alcohol Mouthwash COOL MINT under virtual supervision in the morning. At home, participants will brush and rinse a second time unsupervised daily in the evening and twice daily over weekends and holidays for the first 3 months of the study (up to visit 3). After visit 3, for the next three months until the end of the study, weekday virtual visits will drop to three times a week. First product use will occur at the site under supervision. Participants will be required to record their daily product use times on a participant diary.
  Interventions: Drug: Colgate Cavity Protection Toothpaste; Drug: LISTERINE ZERO Alcohol Mouthwash COOL MINT
- Interdental Brush/Brush (Experimental): Participants will use their interdental brush according to their personalized "mouth map", rinse with water then brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protections Toothpaste for 2 timed minutes under virtual supervision in the morning. At home, participants will brush a second time unsupervised daily in the evening and twice daily over weekends and holidays for the first 3 months of the study (up to visit 3). After visit 3, for the next three months until the end of the study, weekday virtual visits will drop to three times a week. Throughout the study, only tooth brushing will be performed a second time in the evening (no interdental brush use). First product use will occur at the site under supervision. Participants will be required to record their daily product use times on a participant diary.
  Interventions: Drug: Colgate Cavity Protection Toothpaste; Device: TePe Original Interdental Brush
- Interdental Brush/Brush/Rinse (LISTERINE COOL MINT Antiseptic Mouthwash) (Experimental): Participants will use their interdental brush according to their personalized "mouth map," rinse with water, brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protections Toothpaste for 2 timed minutes and then rinse for 30 seconds with LISTERINE COOL MINT Antiseptic Mouthwash under virtual supervision in the morning. At home, participants will brush and rinse a second time unsupervised daily in the evening and twice daily over weekends and holidays for the first 3 months of the study (up to visit 3). After visit 3, for the next three months until the end of the study, weekday virtual visits will drop to three times a week. Throughout the study, only tooth brushing will be performed a second time in the evening (no interdental brush use). First product use will occur at the site under supervision. Participants will be required to record their daily product use times on a participant diary.
  Interventions: Drug: Colgate Cavity Protection Toothpaste; Drug: LISTERINE COOL MINT Antiseptic Mouthwash; Device: TePe Original Interdental Brush
- Interdental Brush/Brush/Rinse (LISTERINE ZERO Alcohol Mouthwash COOL MINT) (Experimental): Participants will use their interdental brush according to their personalized "mouth map," rinse with water, brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protections Toothpaste for 2 timed minutes and then rinse for 30 seconds with LISTERINEZERO Alcohol Mouthwash COOL MINT under virtual supervision in the morning. At home, participants will brush and rinse a second time unsupervised daily in the evening and twice daily over weekends and holidays for the first 3 months of the study (up to visit 3). After visit 3, for the next three months until the end of the study, weekday virtual visits will drop to three times a week. Throughout the study, only tooth brushing will be performed a second time in the evening (no interdental brush use). First product use will occur at the site under supervision. Participants will be required to record their daily product use times on a participant diary.
  Interventions: Drug: Colgate Cavity Protection Toothpaste; Drug: LISTERINE ZERO Alcohol Mouthwash COOL MINT; Device: TePe Original Interdental Brush

INTERVENTIONS:
Drug: Colgate Cavity Protection Toothpaste — Participants will use Colgate Cavity Protection Toothpaste for brushing teeth twice daily.
Drug: LISTERINE ZERO Alcohol Mouthwash COOL MINT — Participants will use LISTERINE ZERO Alcohol Mouthwash COOL MINT for 30 second after brushing teeth twice daily.
  Arms: Brush/Rinse (LISTERINE ZERO Alcohol Mouthwash COOL MINT); Interdental Brush/Brush/Rinse (LISTERINE ZERO Alcohol Mouthwash COOL MINT)
Drug: LISTERINE COOL MINT Antiseptic Mouthwash — Participants will use LISTERINE COOL MINT Antiseptic Mouthwash for 30 second after brushing teeth twice daily.
  Arms: Interdental Brush/Brush/Rinse (LISTERINE COOL MINT Antiseptic Mouthwash)
Device: TePe Original Interdental Brush — Participants will use Interdental Brush according to their personalized mouth map once daily in the morning.
  Arms: Interdental Brush/Brush; Interdental Brush/Brush/Rinse (LISTERINE COOL MINT Antiseptic Mouthwash); Interdental Brush/Brush/Rinse (LISTERINE ZERO Alcohol Mouthwash COOL MINT)

SUMMARY:
The purpose of this study is to assess the relative effectiveness of oral (mouth) care regimens for the avoidance and treatment of plaque and gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and follow the requirements and restrictions of the study (including willingness to use the assigned study products per instructions, availability on scheduled visit dates and likeliness of completing the clinical study) based upon research site personnel's assessment
* Evidence of a personally signed and dated informed consent document indicating the participant has been informed of all pertinent aspects of the trial
* Able to read and understand (participants capable of reading the documents)
* Able to schedule once daily virtual session during weekdays during the first three months of the study (up to visit 3) and then three times a week for the remainder of the study for interdental brush use and rinsing in real time via a platform such as Zoom, Facetime, Google Meet, Etcetera (etc)
* Adequate oral hygiene (that is, brush teeth daily and exhibit no signs or oral neglect)
* Males and females in good general and oral health without any known allergy to commercial dental products or cosmetics
* Evidence of being fully vaccinated for corona virus disease-2019 (COVID-19) (adults 60 years and older)
* Negative pregnancy urine tests (females of childbearing potential only)
* Females of childbearing potential must be using a medically-acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the study
* A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count
* Participants should have a minimum of 20 interproximal areas where interdental brushes can be inserted
* All interproximal sites must be able to accommodate an interdental brush
* A minimum of 10 percent (%) bleeding sites based on the expanded bleeding index (BI)
* Participants will have evidence of some gingivitis (mild to severe); there will be no minimum or maximum mean Modified Gingival Index (MGI) score for gingivitis or Turesky Modification of the Quigley Hein Plaque Index (TPI) score for plaque
* No more than 3 sites having pocket depths of 5 millimeters (mm) and no sites that are greater than 5 mm in depth
* Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator
* Absence of advanced periodontitis based on a clinical examination at baseline and discretion of the dental examiner
* Absence of dental implants, fixed or removable orthodontic appliance or removable partial dentures or other appliances which may interfere with supervised interdental brushing

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouth rinses and red food dye; Known allergy or sensitivity or history of significant adverse effects to any of the investigational product and/or product ingredients or other ingredients in the products
* Dental prophylaxis within four weeks prior to baseline visit
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* Use of antibiotics, anti-inflammatory or anticoagulant therapy during the study or within the one month prior to the Baseline exam. Intermittent use of certain anti-inflammatory medication is acceptable at the discretion of the investigator
* Use of chemotherapeutic anti-plaque/anti-gingivitis products such as triclosan, essential oils, cetylpyridinium chloride, stannous fluoride or chlorhexidine containing mouthwashes and toothpastes within four weeks prior to baseline
* Regular consumption of probiotic drinks/supplements within one week prior to screening/baseline;
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results)
* Self-reported smokeless tobacco user including snuff, chewing tobacco, vaping and e-cigarette usage
* Suspected alcohol or substance abuse (example, amphetamines, benzodiazepines, cocaine, marijuana, opiates)
* Significant unstable or uncontrolled medical condition which may interfere with a participant's participation in the study, including cancer, chronic kidney disease, chronic obstructive pulmonary disease (COPD), immunocompromised state (weakened immune system) from solid organ transplant, serious heart conditions, (such as heart failure, coronary artery disease, or cardiomyopathies) sickle cell disease, Type 1 or 2 diabetes mellitus)
* Participation in any clinical trial within 30 days of baseline visit
* Participants who were previously screened and ineligible or were randomized to receive investigational product
* Participants who are related to those persons involved directly or indirectly with the conduct of this study (that is, principal investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the participant inappropriate for entry into this study
* COVID-19 restrictions: Participants who fail to meet the criteria of the site's screening consent for preventing Infection in the site's COVID-19 consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Interproximal Mean Turesky Plaque Index (TPI) After 24 Weeks of Product Use | After 24 weeks of product use
  Interproximal mean TPI after 24 weeks of product use will be reported. Plaque area will be scored by the Turesky Modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (no plaque); 1 (separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (thin, up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (band of plaque wider than 1mm but less than1/3 of the surface); 4 (plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (plaque covering 2/3 or more of the surface).
Interproximal Mean Modified Gingival Index (MGI) After 24 Weeks of Product Use | After 24 weeks of product use
  Interproximal mean MGI after 24 weeks of product use will be reported. Gingivitis will be assessed by the MGI on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (normal [absence of inflammation]), 1 (mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (mild inflammation of the entire gingival unit); 3 (moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).

SECONDARY OUTCOMES:
Interproximal Mean TPI after 4 and 12 Weeks | After 4 and 12 weeks
  Interproximal mean TPI after 4 and 12 weeks will be reported. Plaque area will be scored by the Turesky Modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (no plaque); 1 (separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (thin, up to 1 mm), continuous band of plaque at the gingival margin); 3 (band of plaque wider than 1mm but less than1/3 of the surface); 4 (plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (plaque covering 2/3 or more of the surface).
Interproximal Mean MGI after 4 and 12 Weeks | After 4 and 12 weeks
  Interproximal mean MGI after 4 and 12 weeks will be reported. Gingivitis will be assessed by the MGI on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (normal [absence of inflammation]), 1 (mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (mild inflammation of the entire gingival unit); 3 (moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Interproximal Mean Expanded Bleeding Index (EBI) After 4, 12 and 24 Weeks | After 4, 12 and 24 weeks
  Interproximal mean EBI after 4, 12 and 24 weeks will be reported. Bleeding will be assessed according to the EBI, 168 sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (absence of bleeding after 30 seconds); 1 (bleeding after 30 seconds); 2 (immediate bleeding).
Interproximal Percent Bleeding Sites based on EBI After 4, 12 and 24 Weeks | After 4, 12 and 24 weeks
  Interproximal percent bleeding sites based on EBI after 4, 12 and 24 weeks will be reported. Bleeding will be assessed according to the EBI, 168 Sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (absence of bleeding after 30 seconds); 1 (bleeding after 30 seconds); 2 (immediate bleeding).
Whole Mouth Mean TPI After 4, 12 and 24 Weeks | After 4, 12 and 24 weeks
  Whole mouth mean TPI after 4, 12 and 24 weeks will be reported. Plaque area will be scored by the Turesky Modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (no plaque); 1 (separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (thin, up to 1 mm), continuous band of plaque at the gingival margin); 3 (band of plaque wider than 1mm but less than1/3 of the surface); 4 (plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (plaque covering 2/3 or more of the surface).
Whole Mouth Mean MGI After 4, 12 and 24 Weeks | After 4, 12 and 24 weeks
  Whole mouth mean MGI after 4, 12 and 24 weeks will be reported. Gingivitis will be assessed by the MGI on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (normal [absence of inflammation]), 1 (mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (mild inflammation of the entire gingival unit); 3 (moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole Mouth Mean EBI After 4, 12 and 24 Weeks | After 4, 12 and 24 weeks
  Whole mouth mean EBI after 4, 12 and 24 weeks will be reported. Bleeding will be assessed according to the EBI, 168 Sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (absence of bleeding after 30 seconds); 1 (bleeding after 30 seconds); 2 (immediate bleeding).
Whole Mouth Percent Bleeding Sites based on EBI After 4, 12 and 24 Weeks | After 4, 12 and 24 weeks
  Whole mouth percent bleeding sites based on EBI after 4, 12 and 24 weeks will be reported. Bleeding will be assessed according to the EBI, 168 Sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (absence of bleeding after 30 seconds); 1 (bleeding after 30 seconds); 2 (immediate bleeding).
Marginal Mean TPI After 4, 12 and 24 Weeks | After 4, 12 and 24 weeks
  Marginal mean TPI after 4, 12 and 24 weeks will be reported. Plaque area will be scored by the Turesky Modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (no plaque); 1 (separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (thin, up to 1 mm), continuous band of plaque at the gingival margin); 3 (band of plaque wider than 1mm but less than1/3 of the surface); 4 (plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (plaque covering 2/3 or more of the surface).
Marginal Mean MGI After 4, 12 and 24 Weeks | After 4, 12 and 24 weeks
  Marginal mean MGI after 4, 12 and 24 weeks will be reported. Gingivitis will be assessed by the MGI on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (normal [absence of inflammation]), 1 (mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (mild inflammation of the entire gingival unit); 3 (moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Marginal Mean EBI After 4, 12 and 24 Weeks | After 4, 12 and 24 weeks
  Marginal mean EBI after 4, 12 and 24 weeks will be reported. Bleeding will be assessed according to the EBI, 168 Sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (absence of bleeding after 30 seconds); 1 (bleeding after 30 seconds); 2 (immediate bleeding).
Whole Mouth and Interproximal Mean Pocket Depth After 12 and 24 Weeks | After 12 and 24 weeks
  Whole mouth and interproximal mean pocket depth after 12 and 24 weeks will be reported.
Whole Mouth and Interproximal Mean Bleeding Upon Probing Pocket Depths After 12 and 24 Weeks | After 12 and 24 weeks
  Whole mouth and interproximal mean bleeding upon probing pocket depths after 12 and 24 weeks will be reported. At each of the 6 sites (disto-facial, mid facial, mesio-facial, mesio-lingual, mid-lingual and disto-lingual), bleeding will be observed and scores as: 0=no bleeding and 1=bleeding.
Whole-mouth Mean Rustogi Modified Navy Plaque Index (RMNPI) | Up to 24 weeks
  Whole-mouth mean RMNPI will be reported. Supragingival plaque levels on the facial and lingual surfaces of all scorable teeth will be assessed according to the RMNPI. The facial and lingual surfaces will be divided into nine unequal segments (A, B, C, D, E, F, G, H and I) for a total of 18 sites per tooth that will be scored from 0 to 1, where 0=no plaque and 1=plaque present in the measured segment of the tooth.
Interproximal Mean RMNPI (Sites D and F) | Up to 24 weeks
  Interproximal mean RMNPI (sites D and F) will be reported. Supragingival plaque levels on the facial and lingual surfaces of all scorable teeth will be assessed according to the RMNPI. The facial and lingual surfaces will be divided into nine unequal segments (A, B, C, D, E, F, G, H and I) for a total of 18 sites per tooth that will be scored from 0 to 1, where 0=no plaque and 1=plaque present in the measured segment of the tooth.
Expanded Interproximal Mean RMNPI (Sites D, F, A, and C) | Up to 24 weeks
  Expanded interproximal mean RMNPI (Sites D, F, A, and C) will be reported. Supragingival plaque levels on the facial and lingual surfaces of all scorable teeth will be assessed according to the RMNPI. The facial and lingual surfaces will be divided into nine unequal segments (A, B, C, D, E, F, G, H and I) for a total of 18 sites per tooth that will be scored 0 to 1 where 0=no plaque and 1=plaque present in the measured segment of the tooth.
Observed Bacterial Species Richness As Assessed by Next Generation Deoxyribonucleic Acid (DNA) Sequencing | At baseline, Weeks 4, 12 and 24
  Observed bacterial species richness is measured from collected plaque specimens using Next-Generation DNA sequencing and counting the number of distinct bacterial species. Lower numbers represent scarcity of bacterial types while higher numbers represent large biodiversity of bacterial types detected in collected specimens.
Shannon-Weaver Diversity Index | At baseline, Weeks 4, 12 and 24
  The Shannon-Weaver diversity index will be reported for supragingival plaque assessment.
Total Species Microbial Load | At baseline, Weeks 4, 12 and 24
  Total species microbial load will be reported for supragingival plaque assessment.
Categorical Species Microbial Load | At baseline, Weeks 4, 12 and 24
  Categorical species microbial load will be reported for supragingival plaque assessment.
Individual Species Microbial Load | At baseline, Weeks 4, 12 and 24
  Individual species microbial load will be reported for supragingival plaque assessment.
Sample Clustering Analysis for Composition Change | At baseline, Weeks 4, 12 and 24
  Sample clustering analysis for composition change will be reported for supragingival plaque assessment.
Number of Total Bacteria and Select Species of Interest Expressed in Log10 | At Baseline and Week 24
  Quantification of live total bacteria and select species of interest in supra and sub-gingival plaque using viability quantitative polymerase chain reaction (qPCR) will be reported in Log10 bacterial cell number.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Bauroth K, Charles CH, Mankodi SM, Simmons K, Zhao Q, Kumar LD. The efficacy of an essential oil antiseptic mouthrinse vs. dental floss in controlling interproximal gingivitis: a comparative study. J Am Dent Assoc. 2003 Mar;134(3):359-65. doi: 10.14219/jada.archive.2003.0167. PMID 12699051
- [Background] Sharma N, Charles CH, Lynch MC, Qaqish J, McGuire JA, Galustians JG, Kumar LD. Adjunctive benefit of an essential oil-containing mouthrinse in reducing plaque and gingivitis in patients who brush and floss regularly: a six-month study. J Am Dent Assoc. 2004 Apr;135(4):496-504. doi: 10.14219/jada.archive.2004.0217. PMID 15127875
- [Background] Sharma NC, Charles CH, Qaqish JG, Galustians HJ, Zhao Q, Kumar LD. Comparative effectiveness of an essential oil mouthrinse and dental floss in controlling interproximal gingivitis and plaque. Am J Dent. 2002 Dec;15(6):351-5. PMID 12691269
- [Background] Milleman K, Milleman J, Bosma ML, McGuire JA, Sunkara A, DelSasso A, York T, Cecil AM. Role of Manual Dexterity on Mechanical and Chemotherapeutic Oral Hygiene Regimens. J Dent Hyg. 2022 Jun;96(3):35-45. PMID 35654566
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Background] Van der Weijden GA, Timmerman MF, Nijboer A, Reijerse E, Van der Velden U. Comparison of different approaches to assess bleeding on probing as indicators of gingivitis. J Clin Periodontol. 1994 Oct;21(9):589-94. doi: 10.1111/j.1600-051x.1994.tb00748.x. PMID 7806674
- [Background] Saxton CA, van der Ouderaa FJ. The effect of a dentifrice containing zinc citrate and Triclosan on developing gingivitis. J Periodontal Res. 1989 Jan;24(1):75-80. doi: 10.1111/j.1600-0765.1989.tb00860.x. PMID 2524573
- [Background] CHILTON NW. Studies in the design and analysis of dental experiments. II. A four-way analysis of variance. J Dent Res. 1960 Mar-Apr;39:344-60. doi: 10.1177/00220345600390021601. No abstract available. PMID 13809868
- [Background] Rustogi KN, Curtis JP, Volpe AR, Kemp JH, McCool JJ, Korn LR. Refinement of the Modified Navy Plaque Index to increase plaque scoring efficiency in gumline and interproximal tooth areas. J Clin Dent. 1992;3(Suppl C):C9-12. PMID 1306676
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] 11Newman, MG, Takei, H, Klokkevold, PR, Carranza, FA; 2018; Newman and Carranza's Clinical Periodontology E-Book, 13th Edition; Saunders; p.387.